CLINICAL TRIAL: NCT03464435
Title: A Novel Combined Therapy for Refractory Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOC2017001123
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Refractory Vernal Keratoconjunctivitis; 0.1% tacrolimus; loteprednol etabonate 0.5%/tobramycin 0.3%
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Tacrolimus; Loteprednol Etabonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tacrolimus and loteprednol etabonate/tobramycin (Experimental): topical eye drops
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — All the patients will be treated with 0.1% tacrolimus suspension two times daily, LE/T eye drops four times daily for 1 month. 0.1% tacrolimus will be continued for the last 5 months.
  Other Names: loteprednol etabonate 0.5%/tobramycin 0.3% (LE/T)

SUMMARY:
To evaluate the efficacy and safety of 0.1% tacrolimus combined with loteprednol etabonate 0.5%/tobramycin 0.3% (LE/T) in vernal keratoconjunctivitis (VKC) patients resistant to conventional treatment. This prospective 6-mouth period study aims to include 20 severe VKC patients who were not responding to conventional treatments. All the patients will be treated with 0.1% tacrolimus suspension two times daily, LE/T eye drops four times daily for 1 month. Additionally, 0.1% olopatadine two times daily and preservative-free artificial tears four times daily will be used. After the first month, LE/T will be stopped, with other treatments continued for the last 5 months. Visual acuity and intraocular pressure (IOP) will be measured at enrollment and 1, 2, 3 and 6 months after treatment. Besides, 6 subjective symptoms and 6 clinical signs will be graded at each visit based on a 4-point scale. The primary endpoints are the change in symptoms and objective signs. Treatment failure will be recorded if extra corticosteroids were required.

ELIGIBILITY:
Inclusion Criteria:

* vernal keratoconjunctivitis patients resistant to conventional treatments

Exclusion Criteria:

* Patients diagnosed with other coexisting eye disease; with a confirmed or possible pregnancy; younger than 5 years old; had presence of systemic diseases other than coexisting allergic rhinitis, asthma, and atopic dermatitis; reported hypersensitivity to tacrolimus

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
the change of objective ocular signs | before treatment and 1, 2, 3 and 6 months after treatment
  doctors judge the change of conjunctival injection, conjunctival edema, papillae, cobblestone papillae, limbal inflammation and corneal epithelial staining

SECONDARY OUTCOMES:
the change of Best corrected visual acuity | before treatment and 1, 2, 3 and 6 months after treatment
  doctors measure the change of BCVA
the change of intraocular pressure | before treatment and 1, 2, 3 and 6 months after treatment
  doctors measure the change of BCVA
the change of subjective ocular symptoms | before treatment and 1, 2, 3 and 6 months after treatment
  patients report the change of itching, redness, burning, photophobia, grittiness, and mucus discharge